CLINICAL TRIAL: NCT02580786
Title: Breastfeeding Preterm Infants - The Efficacy of Internet-based Peer Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Hannakaisa Niela-Vilen, MNSc, Doctoral candidate, University of Turku
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 26/2011
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Breast Feeding; Infant, Premature
MeSH Terms: conditions — Breast Feeding; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breastfeeding peer support (Experimental): Internet-based breastfeeding peer-support group in social media (Facebook). The mothers are allowed to use the group based on their individual needs from the recruitment to the first birthday of their child. Peer support is provided by three voluntary mothers. The mothers can discuss breastfeeding-related issues and ask questions. A midwife will moderate the group.
  Interventions: Behavioral: Breastfeeding peer support
- Routine breastfeeding support (No Intervention): Routine breastfeeding support provided in the hospital and in the maternal and child health clinics

INTERVENTIONS:
Behavioral: Breastfeeding peer support
  Arms: Breastfeeding peer support

SUMMARY:
This study examines if the internet-based peer support has an effect on the breastfeeding attitude or the duration of breastfeeding in preterm infants and their mothers compared with mothers with routine care. The factors associated with the initiation of breastfeeding in the neonatal intensive care unit will be determined. In addition, the perceptions of the mothers of preterm infants about their needs and problems when breastfeeding their preterm infants are described.

ELIGIBILITY:
Inclusion Criteria:

* Mothers giving birth before full 35 gestational weeks in a study hospital

Exclusion Criteria:

* The mother not able to speak Finnish
* The infant's condition is critical (based on the paediatrician),
* The mother has a syndrome or illness preventing breastfeeding

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Duration of breastfeeding | 12 months
Breastfeeding attitude with Iowa Infant Feeding Attitude Scale | 6 months
  Iowa Infant Feeding Attitude Scale (IIFAS) is used to measure breastfeeding attitude

SECONDARY OUTCOMES:
Initiation of breastfeeding (postnatal age of the preterm infant) | 2 months
  The postnatal age (days), when the preterm infant initiates breastfeeding for the first time, is measured
Duration of expressing milk | 12 months